CLINICAL TRIAL: NCT04260269
Title: Feasibility of Switching Fluoropyrimidine Due to Cardiotoxicity in Patients with Solid Tumors: a Retrospective, International and Non-interventional Study
Brief Title: Feasibility of Switching Fluoropyrimidine Due to Cardiotoxicity Study
Acronym: CardioSwitch
Status: Enrolling by invitation | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Pia Osterlund, Associate Professor Oncology, Tampere University Hospital
Other Study IDs: R18045
Record Dates: First submitted 2020-01-22; First posted 2020-02-07 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor
MeSH Terms: interventions — S 1 (combination); tegafur-gimeracil-oteracil; Capecitabine; Fluorouracil; Tegafur; trifluridine tipiracil drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Fluoropyrimidine — This is the assessment of a specific evaluation of cardiac safety for patients with solid tumors who have experienced cardiotoxicity grade 1-4 during treatment with a fluoropyrimidine based treatment and are re-challenged with a different fluoropyrimidine.
  This multicentre, retrospective database is built to assess the impact on the cardiac and global safety of two different fluoropyrimidine based treatment regimens, of which the first has caused cardiotoxicity grade 1-4.
  Cardiac data will be collected by medical record review from initiation of first fluoropyrimidine-based treatment and switch to second fluoropyrimidine-based treatment until death or last follow-up. Basic demographics, cancer and treatment information from the whole course of cancer until death or last follow-up.
  Other Names: S-1 / Teysuno; capecitabine; 5-fluorouracil; tegafur; trifluridine-tipiracil / Lonsurf

SUMMARY:
The purpose of the present study is to evaluate cardiotoxicity during re-challenge of a different modality of fluoropyrimidine (primary end-point S-1 and secondary any other fluoropyrimidine) after having perceived cardiotoxicity with a fluoropyrimidine based regimen previously. The patient population is being treated for solid tumors.

DETAILED DESCRIPTION:
Fluoropyrimidine chemotherapy agents, such as 5-fluorouracil and capecitabine, are occasionally associated with cardiotoxicity that may manifest as chest pain, ECG alterations, cardiac arrhythmia, and rarely myocardial infarction and sudden death. Clinical fluoropyrimidine cardiotoxicity is infrequent (1-8% of patients), but subclinical toxicity may be much more common (up to one third of patients). The underlying mechanisms are not well understood, but they may include abnormal coronary artery contractility or spasm, and myocardial toxicity. Cardiotoxicity may be less frequent with S-1 (a combination of tegafur, gimeracil and oteracil at a molar ratio of 1:0.4:1) as compared with 5-fluorouracil and capecitabine, but head-to-head comparisons are lacking.

Anecdotal evidence suggests that patients who have cardiotoxicity on other fluoropyrimidines may be successfully treated with S-1. The purpose of this retrospective study is to compare different 5-fluorouracil-based dosing modalities and S-1, and compare cardiotoxicity during these treatments.

The patient population was treated for solid tumors with a 5-fluorouracil based regimen and had a cardiac event grade 1-4. All patients were re-challenged with a different fluoropyrimidine or S-1 and assessed for cardiotoxicity during re-challenge.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor
* Cardiotoxicity grade 1-4 during fluoropyrimidine-based treatment
* Re-challenge with a different fluoropyrimidine-based therapy

Exclusion Criteria:

• Participation in a trial with experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who fulfil the following inclusion criteria will be included in the database until the target number of patients has been included:
  * Solid tumor
  * Cardiotoxicity grade 1-4 during fluoropyrimidine-based treatment
  * Re-challenge with a different fluoropyrimidine-based treatment. Primary endpoint is switch to S-1 and secondary any fluoropyrimidine population.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of fluoropyrimidine related cardiac toxicity after switch to S-1 based treatment | After switch to and during one line of S-1 based chemotherapy (average 6 months)
  Cardiac tolerability according to NCI-CTCAE following cardiotoxicity initiated switch of fluoropyrimidine to S-1

SECONDARY OUTCOMES:
Recurrence of fluoropyrimidine related cardiac toxicity after switch to any fluoropyrimidine | After switch to and during one line of another fluoropyrimidine regimen (average 6 months)
  Cardiac tolerability according to NCI-CTCAE following cardiotoxicity initiated switch of fluoropyrimidine to another fluoropyrimidine chemotherapy
Cardiac symptoms during fluoropyrimidine chemotherapy | During one line of fluoropyrimidine based chemotherapy (average 6 months)
  Frequency and severity according to NCI-CTCAE of cardiac symptoms during different fluoropyrimidines and the correlation with other added cytotoxics or biologics
Diagnostic work-up | During one line of fluoropyrimidine based chemotherapy (average 6 months)
  Diagnostic work-up for cardiotoxicity in real world data
Time-lines for cardiotoxicity | During one line of fluoropyrimidine based chemotherapy (average 6 months)
  Time-lines for appearance of cardiotoxicity during fluoropyrimidine-based chemotherapy
Dose-intensity | During one cycle (average 3 weeks) of fluoropyrimidine-based chemotherapy causing cardiac toxicity
  Dose-intensity of the therapy at the cycle causing cardiotoxicity
Alteration in cardiac functional parameters during fluoropyrimidine treatment induced cardiotoxicity | During one cycle (average 3 weeks) of fluoropyrimidine-based chemotherapy causing cardiac toxicity
  The alterations of (if evaluated), graded as normal, non-significant abnormalities or significant abnormalities.:
  * ECG abnormalities
  * Ejection fraction in %
  * Coronary artery status on angiogram
  * Cardiac arrhythmias in ECG, Holter or cardiac monitor registration
  * Plasma troponin concentration and other cardiac enzymes and other laboratory tests as within reference range ro abnormal
  * Serum alpha-fluoro-beta-alanine (FBAL) concentration

CONTACTS AND LOCATIONS:
Locations (13):
- Odense University Hospital, Odense, Denmark
- Finland (4):
  - Department of Oncology, Tampere, Pirkanmaa
  - Helsinki University Central Hospital, Helsinki, Uusimaa
  - Oulu university hospital, Oulu
  - Turku university hospital, Turku
- Landspitali, Reykjavik, Iceland
- St. Vincents University Hospital, Dublin, Ireland
- Academic Medical Center, Amsterdam, Netherlands
- Haukeland University Hospital, Bergen, Norway
- Sweden (4):
  - Skone university hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Sundsvall hospital, Sundsvall
  - Uppsala academic hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwakman JJM, Baars A, van Zweeden AA, de Mol P, Koopman M, Kok WEM, Punt CJA. Case series of patients treated with the oral fluoropyrimidine S-1 after capecitabine-induced coronary artery vasospasm. Eur J Cancer. 2017 Aug;81:130-134. doi: 10.1016/j.ejca.2017.05.022. Epub 2017 Jun 15. No abstract available. PMID 28623776
- [Background] Kwakman JJ, Simkens LH, Mol L, Kok WE, Koopman M, Punt CJ. Incidence of capecitabine-related cardiotoxicity in different treatment schedules of metastatic colorectal cancer: A retrospective analysis of the CAIRO studies of the Dutch Colorectal Cancer Group. Eur J Cancer. 2017 May;76:93-99. doi: 10.1016/j.ejca.2017.02.009. Epub 2017 Mar 10. PMID 28286287
- [Background] Winther SB, Zubcevic K, Qvortrup C, Vestermark LW, Jensen HA, Krogh M, Sorbye H, Pfeiffer P; Academy of Geriatric Cancer Research (AgeCare). Experience with S-1 in older Caucasian patients with metastatic colorectal cancer (mCRC): Findings from an observational chart review. Acta Oncol. 2016 Jul;55(7):881-5. doi: 10.3109/0284186X.2016.1161825. Epub 2016 May 16. PMID 27181284
- [Background] Ye JX, Liu AQ, Ge LY, Zhou SZ, Liang ZG. Effectiveness and safety profile of S-1-based chemotherapy compared with capecitabine-based chemotherapy for advanced gastric and colorectal cancer: A meta-analysis. Exp Ther Med. 2014 May;7(5):1271-1278. doi: 10.3892/etm.2014.1576. Epub 2014 Feb 24. PMID 24940424
- [Background] Yeh ET, Bickford CL. Cardiovascular complications of cancer therapy: incidence, pathogenesis, diagnosis, and management. J Am Coll Cardiol. 2009 Jun 16;53(24):2231-47. doi: 10.1016/j.jacc.2009.02.050. PMID 19520246
- [Background] Deboever G, Hiltrop N, Cool M, Lambrecht G. Alternative treatment options in colorectal cancer patients with 5-fluorouracil- or capecitabine-induced cardiotoxicity. Clin Colorectal Cancer. 2013 Mar;12(1):8-14. doi: 10.1016/j.clcc.2012.09.003. Epub 2012 Oct 26. PMID 23102544
- [Background] Polk A, Vaage-Nilsen M, Vistisen K, Nielsen DL. Cardiotoxicity in cancer patients treated with 5-fluorouracil or capecitabine: a systematic review of incidence, manifestations and predisposing factors. Cancer Treat Rev. 2013 Dec;39(8):974-84. doi: 10.1016/j.ctrv.2013.03.005. Epub 2013 Apr 10. PMID 23582737
- [Derived] Osterlund P, Kinos S, Pfeiffer P, Salminen T, Kwakman JJM, Frodin JE, Shah CH, Sorbye H, Ristamaki R, Halonen P, Soveri LM, Heerva E, Algars A, Barlund M, Hagman H, McDermott R, O'Reilly M, Rockert R, Liposits G, Kallio R, Flygare P, Teske AJ, van Werkhoven E, Punt CJA, Glimelius B. Continuation of fluoropyrimidine treatment with S-1 after cardiotoxicity on capecitabine- or 5-fluorouracil-based therapy in patients with solid tumours: a multicentre retrospective observational cohort study. ESMO Open. 2022 Jun;7(3):100427. doi: 10.1016/j.esmoop.2022.100427. Epub 2022 Mar 30. PMID 35798468